CLINICAL TRIAL: NCT06863272
Title: MK-2400-01A Substudy: A Phase 1/2, Open-label Umbrella Substudy of MK-2400-U01 Master Protocol to Evaluate the Safety and Efficacy of Ifinatamab Deruxtecan-based Treatment Combinations or Ifinatamab Deruxtecan Alone in Participants With Metastatic Castration-resistant Prostate Cancer (mCRPC) (IDeate-Prostate02)
Brief Title: A Clinical Study of Ifinatamab Deruxtecan Based Treatment Combinations or as Monotherapy to Treat Metastatic Castrate Resistant Prostate Cancer (mCRPC) (MK-2400-01A/IDeate-Prostate02)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2400-01A; MK-2400-01A (Other: MSD); 2024-516036-94-00 (Registry Identifier: EU CT); U1111-1310-5406 (Registry Identifier: UTN); IDeate-Prostate02 (Other: MSD)
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Castration-Resistant Prostatic Cancer; Metastasis
MeSH Terms: conditions — Prostatic Neoplasms, Castration-Resistant; Neoplasm Metastasis | interventions — Docetaxel; abiraterone; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Docetaxel (Active Comparator): Participants will receive docetaxel at a determined dose every 3 weeks (Q3W) for a maximum of 10 cycles. Each cycle is 21 days.
  Interventions: Drug: Docetaxel
- Ifinatamab Deruxtecan (I-DXd) (Experimental): Participants will receive I-DXd at a determined dose Q3W until unacceptable toxicity, progressive disease (PD), death or withdrawal of consent.
  Interventions: Drug: Ifinatamab Deruxtecan; Drug: Rescue Medication
- I-DXd + MK-5684 (Experimental): Following a dose escalation regimen with I-DXd, participants will receive I-DXd at a determined dose until unacceptable toxicity, PD, death or withdrawal of consent PLUS MK-5684 at a determined dose until any of the criterion for discontinuation of study intervention is met.
  Interventions: Drug: Ifinatamab Deruxtecan; Drug: MK-5684; Drug: Rescue Medication
- I-DXd +ARPI (Abiraterone or Enzalutamide) (Experimental): Following a dose escalation regimen with I-DXd, participants will receive I-DXd at a determined dose until unacceptable toxicity, PD, death or withdrawal of consent PLUS ARPI (Androgen Receptor Pathway Inhibitor) - Abiraterone acetate OR Enzalutamide at a determined dose until any of the criterion for discontinuation of study intervention is met.
  Interventions: Drug: Ifinatamab Deruxtecan; Drug: Abiraterone; Drug: Enzalutamide; Drug: Rescue Medication

INTERVENTIONS:
Drug: Docetaxel — Administered via Intravenous (IV) infusion at a specified dose on specified days
  Arms: Docetaxel
Drug: Ifinatamab Deruxtecan — Administered via IV infusion at a specified dose on specified days
  Other Names: I-DXd, MK-2400, DS-7300a
  Arms: I-DXd + MK-5684; I-DXd +ARPI (Abiraterone or Enzalutamide); Ifinatamab Deruxtecan (I-DXd)
Drug: MK-5684 — Administered orally at a specified dose on specified days
  Other Names: ODM-208
  Arms: I-DXd + MK-5684
Drug: Abiraterone — Administered orally at a specified dose on specified days
  Arms: I-DXd +ARPI (Abiraterone or Enzalutamide)
Drug: Enzalutamide — Administered orally at a specified dose on specified days
  Arms: I-DXd +ARPI (Abiraterone or Enzalutamide)
Drug: Rescue Medication — Before each dose of I-DXd, participants are required to take premedication for prevention of nausea and vomiting with a 2- or 3-drug combination regimen (eg, dexamethasone with either a 5-HT3 receptor antagonist or an NK-1 receptor antagonist as well as other drugs as indicated) per approved product label.
  Arms: I-DXd + MK-5684; I-DXd +ARPI (Abiraterone or Enzalutamide); Ifinatamab Deruxtecan (I-DXd)

SUMMARY:
The purpose of this substudy is to assess the efficacy and safety of ifinatamab deruxtecan (I-DXd), given alone or with other treatments in participants with metastatic castration-resistant prostate cancer (mCRPC). The goals of this study are to learn about:

* The safety of the study treatment and if people tolerate it.
* A safe dose level of I-DXd that can be used with other treatments.
* Participant levels of prostate specific antigen (PSA) during treatment.

DETAILED DESCRIPTION:
This sub study MK-2400-01A assesses treatments for metastatic castration-resistant prostate cancer (mCRPC).

The master screening protocol is MK-2400-U01

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has histologically- or cytologically-confirmed adenocarcinoma of the prostate without small cell histology
* Has prostate cancer progression while on androgen deprivation therapy (ADT) (or post bilateral orchiectomy) within 6 months before Screening
* Has current evidence of metastatic disease
* Has received prior treatment with 1 or 2 androgen receptor pathway inhibitors (ARPIs) and progressed during or after treatment
* Participants receiving bone resorptive therapy (including, but not limited to bisphosphonate or denosumab) must have been on stable doses for ≥4 weeks before allocation/randomization
* An Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 assessed within 10 days before allocation/randomization
* Has prior treatment with poly-ADP-ribose polymerase inhibitors (PARPi) if indicated by local approved regimen or were deemed ineligible to receive PARPi by the investigator

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* History of (non-infectious) interstitial lung disease (ILD)/pneumonitis that required steroids, or has current ILD/pneumonitis or suspected ILD/pneumonitis
* Clinically severe pulmonary compromise resulting from intercurrent pulmonary illnesses
* Uncontrolled or significant cardiovascular disease
* History of pituitary dysfunction
* Poorly controlled diabetes mellitus
* History or current condition of adrenal insufficiency (eg, Addison's disease)
* Has received prior treatment with taxane-based chemotherapy agent for metastatic castration-resistant prostate cancer (mCRPC).
* Chronic steroid treatment (dose of >10 mg daily prednisone equivalent), except for low-dose inhaled steroids (for asthma/chronic obstructive pulmonary disease), topical steroids (for mild skin conditions), or intra-articular steroid injections
* Received prior radiotherapy within 2 weeks of start of study intervention, or has radiation-related toxicities, requiring corticosteroids
* Known additional malignancy that is progressing or has required active treatment within the past 3 years
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Active autoimmune disease that has required systemic treatment in the past 2 years
* History of allogeneic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-07-03 (Actual); Primary Completion 2030-02-18 (Estimated); Study Completion 2030-02-24 (Estimated)

PRIMARY OUTCOMES:
Efficacy Phase: Number of Participants Who Experience One or More Dose-Limiting Toxicities (DLTs) - Combination Arms Only | Up to approximately 21 days
  The following events if considered drug related by the Investigator, will be considered a DLT: Grade 4 nonhematologic toxicity (not based on laboratory value); Grade 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia; Grade 4 thrombocytopenia of any duration; Grade 3 thrombocytopenia associated with clinically significant bleeding; Nonhematologic AEs ≥Grade 3 with exceptions; Grade 3 or Grade 4 non-hematologic laboratory values if requires medical intervention, leads to hospitalization, persists for >1 week, or results in a Drug-induced Liver Injury with exceptions; Grade 3 or 4 febrile neutropenia; Study intervention - related toxicities that lead to discontinuation of study treatment during Cycle 1; Prolonged delay (>2 weeks) in initiating Cycles 2 due to treatment-related toxicity; Missing >25% of study intervention doses as a result of treatment-related AE during Cycle 1; Grade 5 toxicity.
Efficacy Phase: Number of Participants Who Experienced an Adverse Event (AE) | Up to approximately 54 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Efficacy Phase: Number of Participants Who Discontinued Study Intervention Due to an AE | Up to approximately 24 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Efficacy Phase: Prostate-Specific Antigen (PSA) response rate | Up to approximately 54 months
  PSA response is defined per prostate cancer working group (PCWG) criteria as a reduction in the PSA level of 50% or more from baseline measured at consecutive assessments at least 3 weeks apart.
Safety Lead-in Phase: Number of Participants Who Experience One or More Dose-Limiting Toxicities (DLTs) - Combination Arms Only | Up to approximately 21 days
  The following events if considered drug related by the Investigator, will be considered a DLT: Grade 4 nonhematologic toxicity (not based on laboratory value); Grade 4 hematologic toxicity lasting ≥7 days, except thrombocytopenia; Grade 4 thrombocytopenia of any duration; Grade 3 thrombocytopenia associated with clinically significant bleeding; Nonhematologic AEs ≥Grade 3 with exceptions; Grade 3 or Grade 4 non-hematologic laboratory values if requires medical intervention, leads to hospitalization, persists for >1 week, or results in a Drug-induced Liver Injury with exceptions; Grade 3 or 4 febrile neutropenia; Study intervention - related toxicities that lead to discontinuation of study treatment during Cycle 1; Prolonged delay (>2 weeks) in initiating Cycles 2 due to treatment-related toxicity; Missing >25% of study intervention doses as a result of treatment-related AE during Cycle 1; Grade 5 toxicity.
Safety Lead-in Phase: Number of Participants Who Experienced an Adverse Event (AE) - Combination Arms Only | Up to approximately 21 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Safety Lead-in Phase: Number of Participants Who Discontinued Study Intervention Due to an AE - Combination Arms Only | Up to approximately 21 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 54 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per PCWG-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1). The percentage of participants who experience CR or PR as assessed by Blinded Independent Central Review (BICR) will be presented.
Radiographic Progression-Free Survival (rPFS) | Up to approximately 54 months
  rPFS is defined as the time from randomization to the first documented progressive disease (PD) per PCWG-modified RECIST 1.1 based on BICR or death due to any cause, whichever occurred first. Per PCWG-modified RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions or ≥2 new bone lesions was also considered PD. PCWG-modified RECIST is similar to RECIST 1.1 with the exception that a confirmation assessment of PD (>4 weeks after the initial PD) is required for participants who remain on treatment following a documented PD per RECIST 1.1 and PCWG rules include new bone lesions. The rPFS per PCWG-modified RECIST as assessed by BICR for all participants is presented. The nonparametric Kaplan-Meier method will be used to estimate the rPFS curve in each treatment arm
Overall Survival (OS) | Up to approximately 54 months
  Overall survival (OS) is defined as the time from randomization to death due to any cause. The nonparametric Kaplan-Meier method will be used to estimate the survival curves.
Duration of Response (DOR) | Up to approximately 54 months
  DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per PCWG-modified RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of ≥ 2 new bone lesions is also considered PD. DOR as assessed by BICR is presented. The nonparametric Kaplan-Meier method will be used to estimate the DOR in each treatment arm.
Time from allocation/randomization to initiation of the first subsequent anticancer therapy (TFST) | Up to approximately 54 months
  TFST is defined as the time from randomization to initiation of the first subsequent anticancer therapy or death, whichever occurs first. The nonparametric Kaplan-Meier method will be used to estimate the TFST in each treatment arm.
Time to Prostate-Specific Antigen (PSA) Progression | Up to approximately 54 months
  Time to PSA progression is defined as the time from randomization to PSA progression. Participants without PSA progression will be censored at the last PSA assessment date. The PSA progression date is defined as the date of:
  1) ≥25% increase and ≥2 ng/mL above the nadir, confirmed by a second value ≥3 weeks later if there is PSA decline from baseline, OR 2) ≥25% increase and ≥2 ng/mL increase from baseline beyond 12 weeks if there is no PSA decline from baseline.
Time to pain progression (TTPP) | Up to approximately 54 months
  The time from allocation/randomization to pain progression based on the Brief Pain Inventory-Short Form (BPI-SF) Item 3 "worst pain in 24 hours" and by the Analgesic Quantification Algorithm (AQA) score.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (60):
- United States (3):
  - MedStar Georgetown Cancer Institute at MedStar Washington Hospital Center ( Site 0026), Washington D.C., District of Columbia
  - The West Clinic, PLLC dba West Cancer Center ( Site 0005), Germantown, Tennessee
  - Fred Hutchinson Cancer Center ( Site 0013), Seattle, Washington
- Argentina (2):
  - Instituto Alexander Fleming ( Site 0202), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Fundación CORI para la Investigación y Prevención del Cáncer ( Site 0200), La Rioja
- Macquarie University-MQ Health Clinical Trials Unit ( Site 0801), Macquarie University, New South Wales, Australia
- Brazil (8):
  - Liga Norte Riograndense Contra o Câncer ( Site 0271), Natal, Rio Grande do Norte
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre ( Site 0270), Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento ( Site 0278), Porto Alegre, Rio Grande do Sul
  - Hospital Universitário São Francisco de Assis - Bragança Paulista ( Site 0268), Bragança Paulista, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto ( Site 0263), São José do Rio Preto, São Paulo
  - Hospital Alemao Oswaldo Cruz ( Site 0279), São Paulo, São Paulo
  - IPITEC ( Site 0275), São Paulo
  - IBCC - Instituto Brasileiro de Controle do Câncer ( Site 0269), São Paulo
- Canada (3):
  - BC Cancer - Vancouver Center ( Site 0103), Vancouver, British Columbia
  - Sunnybrook Research Institute ( Site 0109), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0102), Toronto, Ontario
- Chile (4):
  - Clinica Universidad Catolica del Maule ( Site 0236), Talca, Maule Region
  - FALP ( Site 0232), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 0231), Santiago, Region M. de Santiago
  - ONCOCENTRO APYS ( Site 0234), Viña del Mar, Región de Valparaíso
- France (5):
  - Institut Bergonié - Centre Régional de Lutte Contre Le Cancer de Bordeaux et Sud Ouest ( Site 0498), Bordeaux, Gironde
  - Centre Oscar Lambret ( Site 0495), Lille, Nord
  - Institut De Cancerologie De L Ouest ( Site 0494), Saint-Herblain, Pays de la Loire Region
  - Centre Hospitalier de la Côte Basque ( Site 0496), Bayonne, Pyrenees-Atlantiques
  - centre hospitalier lyon sud ( Site 0497), Pierre-Bénite, Rhone
- Germany (3):
  - NCT ( Site 0528), Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Jena ( Site 0525), Jena, Thuringia
  - Universitaetsklinikum Hamburg-Eppendorf ( Site 0524), Hamburg
- Beaumont Hospital, Dublin ( Site 0465), Dublin, Ireland
- Israel (4):
  - Rambam Health Care Campus ( Site 0400), Haifa
  - Rabin Medical Center ( Site 0402), Petah Tikva
  - Sheba Medical Center ( Site 0401), Ramat Gan
  - Sourasky Medical Center ( Site 0403), Tel Aviv
- Italy (5):
  - A.O.U. Federico II di Napoli ( Site 0435), Naples, Napoli
  - AOU San Luigi Gonzaga di Orbassano ( Site 0434), Orbassano, Torino
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia ( Site 0432), Brescia
  - Fondazione IRCCS Istituto Nazionale Dei Tumori ( Site 0431), Milan
  - Fondazione Policlinico Universitario Agostino Gemelli ( Site 0433), Roma
- UMC St. Radboud ( Site 0679), Nijmegen, Gelderland, Netherlands
- Auckland City Hospital ( Site 0831), Auckland, New Zealand
- Poland (4):
  - Uniwersytecki Szpital Kliniczny w Poznaniu ( Site 0590), Poznan, Greater Poland Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - Panstwowy Instytut Badawczy w Warszawie ( Site 0586), Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne ( Site 0588), Gdansk, Pomeranian Voivodeship
  - Szpital Wojewódzki im. M.Kopernika Oddział Onk. Klinicznej z Pododdziałem Chemioterapii Jednodniowej ( Site 0587), Koszalin, West Pomeranian Voivodeship
- South Korea (3):
  - Asan Medical Center ( Site 0925), Songpagu, Seoul
  - Severance Hospital Yonsei University Health System ( Site 0924), Seoul
  - Samsung Medical Center ( Site 0926), Seoul
- Spain (4):
  - Hospital Universitario Ramon y Cajal ( Site 0620), Madrid
  - Hospital Clinico San Carlos ( Site 0618), Madrid
  - Hospital Universitario 12 de Octubre ( Site 0622), Madrid
  - Hospital Universitario Virgen del Rocio ( Site 0619), Seville
- Taiwan (2):
  - Taichung Veterans General Hospital ( Site 0902), Taichung
  - Taipei Veterans General Hospital ( Site 0901), Taipei
- Turkey (Türkiye) (2):
  - Baskent University Dr. Turgut Noyan Research and Training Center ( Site 0650), Adana
  - Hacettepe Universitesi Tip Fakultesi ( Site 0648), Ankara
- United Kingdom (4):
  - Addenbrooke's Hospital ( Site 0747), Cambridge, Cambridgeshire
  - St Bartholomew's Hospital ( Site 0749), London, London, City of
  - Royal Free Hospital ( Site 0743), London, London, City of
  - Royal Marsden Hospital (Sutton) ( Site 0741), London, Surrey

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com